CLINICAL TRIAL: NCT03303105
Title: A Multicenter, Randomized, Open-label Trial Evaluating the Long-term Safety and Tolerability of Subcutaneous Administration of TEV-48125 for the Preventive Treatment of Migraine
Brief Title: Long-term Safety and Tolerability of Subcutaneous Administration of TEV-48125 for the Preventive Treatment of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 406-102-00003; JapicCTI-173726 (Other: Japic)
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEV-48125 (225 mg/1 month) group (Experimental): TEV-48125 will be administered subcutaneously once every 4 weeks for a total of 13 doses (at 225 mg once monthly [except for a loading dose of 675 mg in subjects with CM]).
  Interventions: Drug: TEV-48125
- TEV-48125 (675 mg/3 month) group (Experimental): TEV-48125 will be administered subcutaneously once every 12 weeks for a total of 5 doses (at 675 mg once every 3 months).
  Interventions: Drug: TEV-48125

INTERVENTIONS:
Drug: TEV-48125 — TEV-48125 will be administered subcutaneously once every 4 weeks.
  Arms: TEV-48125 (225 mg/1 month) group
Drug: TEV-48125 — TEV-48125 will be administered subcutaneously once every 12 weeks.
  Arms: TEV-48125 (675 mg/3 month) group

SUMMARY:
To evaluate the long-term safety and tolerability of subcutaneous (SC) administration of TEV-48125 (at 225 mg once monthly [except for a loading dose of 675 mg for CM patients] or at 675 mg every 3 months) for the preventive treatment of Chronic Migraine and Episodic Migraine patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of migraine (according to The International Classification of Headache Disorders, third edition [beta version] criteria) or clinical judgment suggests a migraine diagnosis
* Patient fulfills the criteria for Chronic migraine or Episodic migraine in baseline information collected during the 28 day screening period
* Not using preventive migraine medications for migraine or other medical conditions or using no more than 2 preventive migraine medication for migraine or other medical conditions if the dose and regimen have been stable for at least 2 months prior to giving informed consent.
* Patient demonstrates compliance with the electronic headache diary during the screening period by entry of headache data on a minimum of 24 of 28 days and the entered data is judged appropriate by the investigator.

Exclusion Criteria:

- Hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, or ocular disease considered clinically significant in the judgment of the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Saitama Medical University Hospital, Iruma, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sakai F, Suzuki N, Ning X, Ishida M, Usuki C, Iba K, Isogai Y, Koga N. Long-Term Safety and Tolerability of Fremanezumab for Migraine Preventive Treatment in Japanese Outpatients: A Multicenter, Randomized, Open-Label Study. Drug Saf. 2021 Dec;44(12):1355-1364. doi: 10.1007/s40264-021-01119-2. Epub 2021 Oct 23. PMID 34687446

RESULTS

PARTICIPANT FLOW:
Groups:
- TEV-48125 (225 mg/1 Month) Group: TEV-48125 will be administered subcutaneously once every 4 weeks for a total of 13 doses (at 225 mg once monthly [except for a loading dose of 675 mg in subjects with chronic migraine).
Period: Overall Study
Arm/Group | TEV-48125 (225 mg/1 Month) Group | TEV-48125 (675 mg/3 Month) Group
Started | 25 | 25
Completed | 23 | 21
Not Completed | 2 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEV-48125 (225 mg/1 Month) Group | TEV-48125 (675 mg/3 Month) Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (7.9) | 45.8 (7.0) | 46.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 25 | 25 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: * TEAEs are defined as the AEs that started after trial investigational medicinal product (IMP) treatment. Multiple occurrences of TEAEs are counted once per MedDRA preferred term.
  * Specific AE terms are provided in the Adverse Event section.
Time Frame: Baseline (Day 0) up to follow-up visit (Day 562)
Population: Safety Set (SS): Newly enrolled subjects who received the IMP at least once
Measure: Number; unit: percentage of participants
Arm/Group | TEV-48125 (225 mg/1 Month) Group | TEV-48125 (675 mg/3 Month) Group
Number analyzed (Participants) | 25 | 25
percentage of participants | 92.0 | 88.0

2. Secondary Outcome: Mean Change From Baseline in the Monthly (28 Day) Average Number of Migraine Days
Description: Headache-related efficacy endpoints were derived from headache variables collected using an eDiary. On each day, subjects entered headache data in the electronic headache diary for the previous 24-hour period. Subjects who had experienced headache on the previous day answered questions about the headache (ie, occurrence of headache, duration of headache, maximum severity of headache, presence/absence of associated symptoms, and use of acute headache medications). Overall headache duration was recorded numerically, in hours, as well as number of hours with headache of at least moderate severity. If headache was reported, then headache severity was subjectively rated by the subject as mild, moderate, or severe.
  Subjects also recorded the presence or absence of photophobia, phonophobia, nausea, or vomiting, and the status of use of any acute headache medications.
Time Frame: Baseline, Month 12
Population: Full Analysis set (FAS): Newly enrolled subjects for whom electronic headache diary efficacy assessment data at baseline and after the first dose of IMP were available
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | TEV-48125 (225 mg/1 Month) Group | TEV-48125 (675 mg/3 Month) Group
Number analyzed (Participants) | 23 | 22
days/month | -5.9 (4.3) | -1.6 (5.7)

3. Secondary Outcome: Mean Change From Baseline in the Monthly (28 Day) Average Number of Headache Days of at Least Moderate Severity
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | TEV-48125 (225 mg/1 Month) Group | TEV-48125 (675 mg/3 Month) Group
Number analyzed (Participants) | 23 | 22
days/month | -4.3 (4.1) | -2.1 (4.1)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to follow-up visit (Day 562)
Description: Safety Set (SS): Newly enrolled subjects who received the IMP at least once
Arm/Group | TEV-48125 (225 mg/1 Month) Group | TEV-48125 (675 mg/3 Month) Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 2/25
Other Adverse Events (participants affected / at risk) | 20/25 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEV-48125 (225 mg/1 Month) Group (N=25) | TEV-48125 (675 mg/3 Month) Group (N=25)
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TEV-48125 (225 mg/1 Month) Group (N=25) | TEV-48125 (675 mg/3 Month) Group (N=25)
Injection site pruritus (General disorders) | 2 | 1
Injection site induration (General disorders) | 3 | 2
Injection site erythema (General disorders) | 7 | 5
Injection site pain (General disorders) | 1 | 3
Influenza (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 3 | 1
Oral herpes (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 18 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03303105/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT03303105/SAP_001.pdf